CLINICAL TRIAL: NCT02085642
Title: Investigation of the Use of Acupuncture for the Treatment of Spasticity in Chronic Stroke Participants
Acronym: HHSCSTROKEAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HHSCSTROKEACPILOT1
Record Dates: First submitted 2014-02-19; First posted 2014-03-13 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
Keywords: Stroke; Acupuncture; Gait; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): True acupuncture
  Interventions: Other: Acupuncture
- Sham needle (Sham Comparator): Retractable acupuncture needles will be used. No true transcutaneous needling through the skin
  Interventions: Other: Sham needle

INTERVENTIONS:
Other: Acupuncture — Single disposal needle to be used, 0.02 mm x 25 mm in length
  Arms: Acupuncture
Other: Sham needle — Retractable needle with no skin puncture
  Arms: Sham needle

SUMMARY:
The purpose of this study is to investigate if acupuncture is more effective than sham treatment in reducing lower extremity spasticity, and improving gait speed in the chronic phase of stroke recovery.

DETAILED DESCRIPTION:
Background: Stroke is one of the leading causes of death and disability in Canada. There are approximately 50,000 new cases every year. Stroke victims often experience decreased mobility and significant disability as a result of impaired motor control and velocity-dependent muscle hypertonus (spasticity) in the lower extremity. Over the past 25 years, there has been an increasing interest in the use of acupuncture for the management of stroke-related neurological deficits.

Research questions: Is acupuncture more effective than sham treatment in reducing lower extremity spasticity, and improving gait speed in the chronic phase of stroke recovery?

Methodology

Recruitment: Forty patients will be recruited from the out patient rehabilitation program of a university affiliated teaching hospital.

Group Assignment and Blinding:

The study design is a randomized double blind format. Once identified, interested patients will be screened for eligibility by an intake secretary and randomly assigned to sham (n=20) or acupuncture treatment (n=20) groups using a computer random-number-generation system. Sealed envelopes containing the group assignment will be delivered to acupuncture-trained therapists delivering sham or true acupuncture treatment. Treating therapists' interactions will be standardized to minimize therapist/participant interaction bias Treating therapists will remain blinded to outcome assessment results. Patients will be blinded to the receipt of true acupuncture or sham needles. Outcome measurements will be done by a single assessor who is blinded to the group assignment.

Intervention: Subjects will attend 4 acupuncture treatments sessions within a 3 week period. Needles will be applied to the following acupuncture points: Jiao's foot motor sensory scalp points (2 in total) and 2 additional standardized acupuncture points in the lower legs bilaterally based on Traditional Chinese Medicine (TCM) approach. Treatment needles are pre-sterilized single disposable type, 0.20 mm size and 40 mm in length. The locations of the acupuncture point will be cleaned with alcohol (99%) swab. Needles will be left in place for 20 minutes. In the true acupuncture group, needles will be inserted to a depth at which participants report a tingling sensation (as described De-qi in TCM approach). Subjects randomized to the control group will be treated with retractable needles to avoid transcutaneous insertion at the same acupuncture points.

Outcome Measures: The following outcome measures will be assessed by a blinded assessor. Primary outcome measures:2-minute walk test. Secondary outcome measures: ankle range of motion and self report soft tissue tightness. The outcome measures time frame is set at from baseline to the completion of the intervention period at 3 weeks.

Analysis: Descriptive statistics including mean, standard deviation and frequencies will be used to describe the study participants, as appropriate. Paired t-test will be used for the parametric variables, number of steps per minute, distance on a 2-minute walk test and dorsi-flexion range of motion. Significance is set at p smaller than 0.05. All statistical analysis will be two sided and performed with SPSS (V21).

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients between 55 to 70 years old
* Time from stroke onset 12 months but less than 18 months
* Clinical picture: symptoms of hemiparesis from ischemic or hemorrhage stroke which is confirmed with CAT scan or MRI, stable with vital signs
* Independently ambulatory with/without a walking aid and with/without orthoses for 2 minutes
* Exhibit spastic equinovarus hemiparesis gait on the affected side
* Cognitive function level ≥ 23 with the total score on the MiniMental Status Examination

Exclusion Criteria:

* History of more than one episode of stroke
* Receiving Botox injections for treatment of spasticity
* Medically unstable with life-threatening conditions, epileptic seizures, auto-immune disease, acute or chronic infectious disease

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 2 minute walk test | Baseline to 3 weeks
  Two-minute walk tests (2MWT) - Participants are required to walk continuously for 2 minutes, using their regular aids or orthoses, but with no manual support. The walk will take place over a distance of 10m, and participants will be required to change direction of their own accord. The distance walked in a 2-minute interval will be recorded

SECONDARY OUTCOMES:
Change from baseline in self report ankle tightness | Baseline to 3 weeks
  Participant report outcome measure (PROM) - ankle tightness - a self report outcome measures has been widely used for pain in a format of a 10-point visual analog scale (VAS). Recent studies showed the reliability of the adaption of PROM to cover other clinical outcomes and the re is extensive discussion on minimal detectable clinical improvement. Ankle tightness in Achilles tendon will be recorded as a PROM on a 10-point scale with 0 being no tightness and 10 is the most.
Change from baseline in ankle range of motion | Baseline to 3 weeks
  Participant in sitting position, active and passive ankle dorsi-flexion will be measured by a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Enoch K Ho, MPh, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data at conferences and journals related to stroke and/or physiotherapy/acupuncture

REFERENCES:
- [Background] Wu P, Mills E, Moher D, Seely D. Acupuncture in poststroke rehabilitation: a systematic review and meta-analysis of randomized trials. Stroke. 2010 Apr;41(4):e171-9. doi: 10.1161/STROKEAHA.109.573576. Epub 2010 Feb 18. PMID 20167912
- [Background] Zhong C, Bai L, Dai R, Xue T, Wang H, Feng Y, Liu Z, You Y, Chen S, Tian J. Modulatory effects of acupuncture on resting-state networks: a functional MRI study combining independent component analysis and multivariate Granger causality analysis. J Magn Reson Imaging. 2012 Mar;35(3):572-81. doi: 10.1002/jmri.22887. Epub 2011 Nov 8. PMID 22069078